CLINICAL TRIAL: NCT01346111
Title: Multicenter Study for the Generation of a Score of Comorbidities
Brief Title: Multicenter Study of Generation Comorbidity Score
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, MD, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 1385
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Death
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- generation cohort: Included 5 hospitals from Buenos Aires, Argentina

SUMMARY:
The purpose of the study is to generate and valid a co-morbidity score with updated definitions and suitable for use in Argentina in both public and private settings. These tools would allow us to compare different populations in Argentina adjusting for comorbidities. Also, this would potentially help attending physicians and health administrators.

DETAILED DESCRIPTION:
The investigators will generate a co-morbidity score, perform the score validation and generate an online calculator for the score (open access).

Finally, a score validation for extreme values of score will be performed to ensure representativeness of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult 17 older
* admitted to hospital within 72 hours of admission
* non programed admission

Exclusion Criteria:

* negative to participate
* 72 hs mortality expected
* obstetrics admissions

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults, who were admitted to hospital for a non programme admission, medical or surgical admission
Sampling Method: Probability Sample
Enrollment: 2640 (Actual)
Dates: Start 2009-04; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
generate a co-morbidity score | 12 months follow up
  Generate a co-morbidity score that measures the weight for individuals morbidities with respect to death.

CONTACTS AND LOCATIONS:
Overall Officials: Diego H Giunta, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (5):
- Argentina (5):
  - Hospital Interzonal General de Agudos Piñeyro, Junín, Buenos Aires
  - Hospital Complejo Médico de la Policía Federal Argentina Churruca-Visca, Buenos Aires
  - Hospital General de Agudos Vélez Sarfield, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Lagomaggiore, Mendoza